CLINICAL TRIAL: NCT06314061
Title: The Effect of Continuous Glucose Monitoring With Real-time Alerts on Glycaemic Control in Surgical Patients With Diabetes: A Randomised, Clinical Multicentre Trial
Brief Title: The Effect of Continuous Glucose Monitoring in Surgical Patients With Diabetes.
Acronym: WARD-glucose
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Christian S. Meyhoff (Other)
Collaborators: Rigshospitalet, Denmark (Other); Steno Diabetes Center Copenhagen (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor-Investigator, Christian S. Meyhoff, Professor, head of research, MD, PhD, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WARD-glucose RCT v.2.2
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus; Dysglycemia; Perioperative Complication
Keywords: Diabetes Mellitus; Continuous glucose monitoring; Perioperative medicine; Medical devices
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Parallel, 2-group randomised trial blinded for participants
Who Masked: Participant
Masking Description: Participants will not be alerted of dysglycaemia by the Dexcom G7 application, which will be muted. Thus, the alerts on deviating glucose levels will only be given to the care provider (the nursing staff at the ward)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will wear the CGM-device Dexcom G7, and real-time alerts on dysglycaemia and rapidly increasing or falling glucose levels will alert the nursing staff.
  Interventions: Device: Dexcom G7 Continuous Glucose Monitoring (CGM) System (G7)
- Control group (No Intervention): Participants in the control group will wear a blinded CGM device. The nursing staff will monitor glucose levels with standard care using POC blood glucose measurements.

INTERVENTIONS:
Device: Dexcom G7 Continuous Glucose Monitoring (CGM) System (G7) — A continuous glucose monitor which through a sensor in the skin registers glucose levels every 5 minutes. Glucose levels are shown by connecting the sensor to a mobile device or the Dexcom G7 Receiver where realtime alerts on deviating glucose levels will be sent.
  Other Names: Dexcom G7
  Arms: Intervention group

SUMMARY:
The goal of this randomised controlled trial to investigate the effect of continuous glucose monitoring (CGM) compared to standard point-of-care (POC) blood glucose measurements in surgical patients with diabetes in patients.

The main question it aims to answer is:

• Can the use of the CGM device Dexcom G7 with real-time alerts on dysglycaemia increase the time in range for glucose levels as compared with standard monitoring with point-of-care blood glucose in surgical patients with diabetes?

Participants will be asked to wear a CGM device (Dexcom G7, Dexcom Inc.) during their stay in the hospital. For patients in the intervention group, deviations of glucose levels will provide the nursing staff with alerts. All patients will receive standard care of their diabetes. The CGM device will be worn for up to 10 days or until discharge.

DETAILED DESCRIPTION:
This is a prospective randomised controlled multicentre trial on patients living with diabetes who undergo surgery at Rigshospitalet, Copenhagen University, Bispebjerg and Frederiksberg Hospital, Copenhagen University, and Zealand University Hospital, Køge, Denmark

The study aims to investigate the effect of the CGM-device Dexcom G7 CGM in patients with diabetes undergoing surgery on the diabetic control. The Dexcom G7 provides glucose readings every 5 minutes and can send alerts on dysglycaemia (hypo- and hyperglycaemia) to mobile devices held by the nursing staff.

Patients will wear the CGM before, during and up to 10 days postoperatively.

The study will include 200 patients.

This study is part of an overall project that aims to investigate the use of CGM and continuous wireless monitoring of vital signs in patients with diabetes undergoing major surgery. Using this technology, postoperative complications including dysglycaemia can potentially be detected and treated earlier thus improving the perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Medical history with diabetes mellitus (DM1 or DM2 (insulin-dependent and non-insulin-dependent) requiring antidiabetic drug(s)
* Acute or elective abdominal, orthopaedic, urological, or vascular surgery with estimated duration of surgery >45 minutes
* Expected stay for at least one night in the hospital postoperatively

Exclusion Criteria:

* Local skin symptoms including infection at the posterior aspect of the upper arm that does not allow the sensor to be placed on an unaffected skin area
* Known allergy to the equipment plaster
* Known pregnancy
* Patients with pacemaker or implantable cardioverter defibrillator (ICD) device
* Previous or currently scheduled for pancreatectomy (complete or partial)
* Patients receiving hydroxyurea (these drugs may interfere with CGM readings)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) of CGM glucose levels | Perioperatively
  Time in range (TIR) of CGM glucose levels (6.0-10.0 mmol/l) in minutes per 24 hours after discharge from the post-anaesthesia care unit (PACU) until 10 days postoperative (or until discharge)

SECONDARY OUTCOMES:
Duration of hypoglycaemia | Perioperatively
  Duration of hypoglycaemia (<3.9 mmol/L (<70 mg/dL), assessed by CGM, in minutes per 24 hours after discharge from PACU until 10 days postoperative (or until discharge)
Duration of hyperglycaemia | Perioperatively
  Duration of hyperglycaemia (>10.0 mmol/L (>180 mg/dL), assessed by CGM, in minutes per 24 hours after discharge from PACU until 10 days postoperative (or until discharge)
Number of hypoglycaemia events | Perioperatively
  Number of hypoglycaemia (<3.9 mmol/L (<70 mg/dL) events lasting > 15 minutes per 24 hours after discharge from PACU until 10 days postoperative (or until discharge). Events will be reported as number of events per 24 hours and duration of events (defined from period of first detected deviation until the first reading in a normal glucose level
Number of hyperglycaemia events | Perioperatively
  Number of hyperglycaemia (>10.0 mmol/L (>180 mg/dL) events lasting > 15 minutes per 24 hours after discharge from PACU until 10 days postoperative (or until discharge). Events will be reported as number of events per 24 hours and duration of events (defined from period of first detected deviation until the first reading in a normal glucose level
Complications | 30 days postoperatively
  Severity of complications assessed by the Comprehensive Complication Index (CCI) within 30 days

OTHER OUTCOMES:
Serious adverse events | 30 days postoperatively
  Frequency of any serious adverse event within 30 days, defined as any complication fulfilling the Clavien-Dindo classification of > 2
Serious adverse Device-related events | 30 days postoperatively
  Severe Adverse Device-related Events (SADE) within 30 days
Adverse events | 30 days postoperatively
  Frequency of any adverse events within 30 days
Length of stay | Perioperatively
  Postoperative Length of stay (LOS) in days
Readmission | 6 months postoperatively
  Readmission within 6 months
ICU admission | 6 months postoperatively
  ICU admission within 6 months postoperatively
Days alive and out of hospital | 30 days postoperatively
  Days alive and out of hospital within 30 days
Patient experience | Perioperatively
  Patient experience (semi-structured questionnaire will be carried out in a subset of randomised patients from both groups with the focus on sense of security and patient comfort)
Staff experience | Perioperatively
  Staff experience (semi-structured questionnaire will be carried out during the beginning and towards the end of the trial. It will focus from both groups with the focus on sense of security and patient comfort))

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Meyhoff, MD, PhD, Study Director — University Hospital Bispebjerg and Frederiksberg
Locations (3):
- Denmark (3):
  - Department of Anaesthesiology, Centre for Cancer and Organ Diseases, Rigshospitalet, Copenhagen, The Capital Region of Denmark
  - Department of Anaesthesiology and Intensive Care, Bispebjerg Hospital, Copenhagen, The Capital Region of Denmark
  - Zealand University Hospital, Køge

IPD SHARING:
Plan to Share IPD: No
We do not plan making individual patient data available to researchers outside the study group.